CLINICAL TRIAL: NCT01542879
Title: Development of Radiation Free Whole Body MR Imaging Technique for Staging of Children With Cancer.
Brief Title: Development of Radiation Free Whole Body Magnetic Resonance (MR) Imaging Technique for Staging Children With Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heike E Daldrup-Link (Other)
Responsible Party: Sponsor-Investigator, Heike E Daldrup-Link, Associate Professor of Radiology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-20221; IRB-20221 (Other: Stanford IRB); PEDSVAR0017 (Other: OnCore)
Record Dates: First submitted 2012-02-24; First posted 2012-03-02 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- WB-DW-MR scan (Experimental): simultaneous WB-DW-MR scan and 18-F FDG PET scan
  Interventions: Procedure: WB-DW-MR scan; Procedure: 18-F-FDG PET scan; Drug: Ferumoxytol; Procedure: 18-F-FDG PET/MR scan

INTERVENTIONS:
Procedure: WB-DW-MR scan — WB-DW-MR scans will be obtained on a 3T PET-MR system
  Other Names: Whole Body Diffusion Weighted MR scan
Procedure: 18-F-FDG PET scan
  Other Names: Fludeoxyglucose PET scan
Drug: Ferumoxytol
  Other Names: feraheme
Procedure: 18-F-FDG PET/MR scan

SUMMARY:
A research study on the diagnosis of spread of disease for children who have been diagnosed with solid tumors using a new whole body imaging technique and a new MR contrast agent (ferumoxytol). Standard tests that are used to determine the extent and possible spread of a child's disease include magnetic resonance (MR) imaging, computed tomography (CT), Positron Emission Tomography (PET) as well as bone scanning, and metaiodobenzylguanidine (MIBG) scanning. The purpose of this study is to determine if newer imaging tests referred to as whole body diffusion-weighted MR and whole body PET/MR can detect the extent and spread of the disease as accurately or even better as the standard tests (CT, MR and/or PET/CT). The advantage of the new imaging test is that it is associated with no or significantly reduced radiation exposure compared to standard CT and PET/CT imaging tests. The results of whole body MR and PET/MR will be compared with that of the conventional, standard imaging studies for tumor detecting.

DETAILED DESCRIPTION:
Primary Objective: To compare the sensitivity, specificity and accuracy of WB-DW-MR scans (new technique) with 18F- FDG PET or 18F- FDG PET/CT or 18F- FDG PET/MR scans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a solid extra-cranial tumor like malignant lymphoma or malignant sarcoma and
* Scheduled for or completed a 18F-FDG-PET or 18F-FDG-PET/CT tumor staging procedure.
* There will be no restrictions on prior treatment.
* Very young children who need sedation or anesthesia will be excluded from the study.
* In this pediatric & adult study, the participant or parent/guardian is consented, and the patient when a minor is given an assent form and involved in the discussion as appropriate.

Exclusion Criteria:

* MR-incompatible metal implants,
* need of sedation or claustrophobia.
* Hemosiderosis/hemochromatosis (patients can still be included in 2nd branch without ferumoxytol)
* There will be restrictions regarding use of other Investigational Agents: Pt with iron-overload will not receive Ferumoxytol
* History of allergic reactions to similar compounds will be obtained and patients with a positive history of allergic reaction to iron compounds or other severe allergic reactions.will be excluded from the study.
* Pregnant women and fetuses.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2012-02; Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of sensitivity, specificity and accuracy of WB-DW-MR scans to 18-F FDG PET scans. | The outcome will be measured after image acquisition
  To determine sensitivity and specificity for lesion detection on whole-body scans, the body is divided into 10 anatomical regions, and qualified professionals evaluate each region for the presence or absence of tumor lesions. These results are then compared to the gold standard (established through biopsy and follow-up imaging), allowing for the calculation of true positives, false positives, true negatives, and false negatives for each region. Sensitivity and specificity can then be calculated using these values, providing a measure of the scan's accuracy in detecting lesions across different body areas.

SECONDARY OUTCOMES:
Comparison of sensitivity, specificity and accuracy of Ferumoxytol-enhanced whole-body 18-F FDG PET/MR-scans versus standard clinical Gadolinium-enhanced whole-body 18-F FDG PET/MR-scans. | 2 years
  To determine sensitivity and specificity for lesion detection on whole-body scans, the body is divided into 10 anatomical regions, and qualified professionals evaluate each region for the presence or absence of tumor lesions. These results are then compared to the gold standard (established through biopsy or follow-up imaging), allowing for the calculation of true positives, false positives, true negatives, and false negatives for each region. Sensitivity and specificity can then be calculated using these values, providing a measure of the scan's accuracy in detecting lesions across different body areas.

CONTACTS AND LOCATIONS:
Overall Officials: Heike Daldrup-Link, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Institute, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rashidi A, Baratto L, Theruvath AJ, Greene EB, Jayapal P, Hawk KE, Lu R, Seekins J, Spunt SL, Pribnow A, Daldrup-Link HE. Improved Detection of Bone Metastases in Children and Young Adults with Ferumoxytol-enhanced MRI. Radiol Imaging Cancer. 2023 Mar;5(2):e220080. doi: 10.1148/rycan.220080. PMID 36999999
- [Derived] Theruvath AJ, Siedek F, Yerneni K, Muehe AM, Spunt SL, Pribnow A, Moseley M, Lu Y, Zhao Q, Gulaka P, Chaudhari A, Daldrup-Link HE. Validation of Deep Learning-based Augmentation for Reduced 18F-FDG Dose for PET/MRI in Children and Young Adults with Lymphoma. Radiol Artif Intell. 2021 Oct 6;3(6):e200232. doi: 10.1148/ryai.2021200232. eCollection 2021 Nov. PMID 34870211
- [Derived] Theruvath AJ, Siedek F, Muehe AM, Garcia-Diaz J, Kirchner J, Martin O, Link MP, Spunt S, Pribnow A, Rosenberg J, Herrmann K, Gatidis S, Schafer JF, Moseley M, Umutlu L, Daldrup-Link HE. Therapy Response Assessment of Pediatric Tumors with Whole-Body Diffusion-weighted MRI and FDG PET/MRI. Radiology. 2020 Jul;296(1):143-151. doi: 10.1148/radiol.2020192508. Epub 2020 May 5. PMID 32368961
- [Derived] Klenk C, Gawande R, Uslu L, Khurana A, Qiu D, Quon A, Donig J, Rosenberg J, Luna-Fineman S, Moseley M, Daldrup-Link HE. Ionising radiation-free whole-body MRI versus (18)F-fluorodeoxyglucose PET/CT scans for children and young adults with cancer: a prospective, non-randomised, single-centre study. Lancet Oncol. 2014 Mar;15(3):275-85. doi: 10.1016/S1470-2045(14)70021-X. Epub 2014 Feb 19. PMID 24559803